CLINICAL TRIAL: NCT03418532
Title: A Phase 1b/2, Single-arm, Open-label, Multi-center Study of MP0250 in Combination With Osimertinib in Patients With EGFR-mutated Non-squamous Non-small Cell Lung Cancer (NSCLC) Pretreated With Osimertinib
Brief Title: MP0250 DARPin® Protein Plus Osimertinib in Patients With EGFR-mutated NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP0250-CP202
Record Dates: First submitted 2018-01-10; First posted 2018-02-01 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: EGFR-mutated NSCLC (Disorder)
Keywords: DARPin®protein; MP0250; VEGF; HGF; NSCLC; EGFR mutated; Osimertinib
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: The trial was intended to be a Phase 1/2 trial. Trial was terminated before Phase 2 commenced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): MP0250 DARPin® drug candidate (6 mg/kg or 8 mg/kg or 12 mg/kg, infusion) on day 1 of each 21 day cycle. Osimertinib according to label
  Interventions: Combination Product: MP0250 DARPin® drug candidate, Osimertinib

INTERVENTIONS:
Combination Product: MP0250 DARPin® drug candidate, Osimertinib — Number of Cycles: until progression, unacceptable toxicity or other reasons for withdrawal

SUMMARY:
The purpose of this study is to assess the anti-tumor efficacy, safety, tolerability, pharmacokinetics (PK), immunogenicity and biological activity of the MP0250 DARPin® drug candidate in combination with osimertinib orally once daily (o.d.), when administered to patients with EGFR mutated, advanced, non squamous NSCLC after tumor progression on osimertinib and on or after the most recent therapy.

MP0250 is a multi-DARPin® protein with three specificities, able to simultaneously neutralize the activities of vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF) and also to bind to human serum albumin (HSA) to give an increased plasma half-life and potentially enhanced tumor penetration.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic or unresectable locally advanced non-squamous NSCLC with documented EGFR mutation-positive disease
2. Radiologically documented disease progression on previous osimertinib treatment.
3. Radiologically documented disease progression on or after most recent antitumor therapy.
4. Measurable disease according to RECIST 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 2.
6. Men and women ≥18 years old on the day of signing informed consent.
7. Adequate hematological, hepatic and renal function prior to first dose
8. Serum albumin concentration ≥30 g/L
9. Potassium and magnesium within normal range

Exclusion Criteria:

1. Necrotic tumors or tumors close to large blood vessels that may impose an increased bleeding risk when treated with anti-VEGF agents.
2. Second malignancy that is currently clinically significant or required active intervention during the period of 12 months prior to Screening, except early stage non-melanoma skin cancer treated with curative intent.
3. Known pre-existing interstitial or inflammatory lung disease.
4. Clinical signs of or documented leptomeningeal carcinomatosis. Features such as headache, nuchal rigidity, and photophobia may indicate meningeal involvement.
5. Known brain metastases who are clinically unstable
6. Prohibited anti-NSCLC therapies and not having recovered from related AEs to Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤1
7. Any investigational drug within 28 days prior to study treatment.
8. Current participation in any other interventional clinical study (except survival follow up).
9. Neuropathy as residual toxicity after prior antitumor therapy Grade >2
10. Patients taking medications that have the potential to prolong the QT interval
11. Significant cardiac abnormalities
12. Uncontrolled hypertension
13. Significant risk for bleeding
14. Active or recent thrombolic events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Estimate the objective response rate (ORR) | 6 months
  Tumor response will be assessed based on RECIST 1.1 by using CT or MRI

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) graded according to CTCAE, v4.03. | 15 months
  number of patients with AE/SAE on the base of CTCAE (version 4.03)
progression free survival (PFS) | 12 months
  PFS according to RECIST 1.1
duration of response (DOR) | 9 months
  DOR according to RECIST 1.1
overall survival (OS) | 24 months
  time from the date of first dose of MP0250 until death from any cause or until 1 year for all patients
time to response (TTR) | 4 months
  TTR according to RECIST 1.1
Incidence of anti-drug (MP0250) antibody formation | 15 months
  determined as titer of anti-drug antibodies
pharmacokinetics | 15 months
  half-life
pharmacokinetics | 15 months
  clearance
pharmacokinetics | 15 months
  AUC
pharmacokinetics | 15 months
  Cmax

OTHER OUTCOMES:
biomarkers in tissue | 12 months
  biomarkers associated with response or resistance to MP0250, HGF by IHC
biomarkers in blood | 12 months
  biomarkers associated with response or resistance to MP0250, HGF by ELISA

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Scottsdale Healthcare Hospitals, Scottsdale, Arizona
  - City of Hope - Comprehensive Cancer Center, Duarte, California
  - University of California, San Diego, California
  - UCLA Medical Center, Santa Monica, California
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Duke Cancer Institute, Durham, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas

IPD SHARING:
Plan to Share IPD: No